CLINICAL TRIAL: NCT05982873
Title: Expanded Access to Telisotuzumab Adizutecan
Status: Available | Type: Expanded Access
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: C24-738
Record Dates: First submitted 2023-08-01; First posted 2023-08-09 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-09

CONDITIONS: Solid Tumors
Keywords: Expanded Access; Pre-approval Access; Compassionate Use; Special Access Program; Named Patient Basis; Special Access Scheme

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Telisotuzumab Adizutecan — Intravenous (IV) Infusion

SUMMARY:
This is an expanded access program (EAP) for eligible participants. This program is designed to provide access to telisotuzumab adizutecan prior to approval by the local regulatory agency. Availability will depend on territory eligibility. A medical doctor must decide whether the potential benefit outweighs the risk of receiving an investigational therapy based on the individual patient's medical history and program eligibility criteria.

ELIGIBILITY:
Exclusion Criteria:

* There are other suitable treatment options.
* The participant qualifies for ongoing clinical trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=C24-738